CLINICAL TRIAL: NCT03385187
Title: Prospective Validation Study of a Novel Type IV Home Sleep Apnea Test
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ectosense NV (Industry)
Collaborators: Ziekenhuis Oost-Limburg (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17/034U
Record Dates: First submitted 2017-12-20; First posted 2017-12-28 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-03

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NightOwl HSAT (Other): Patient undergoes a NightOwl sleep apnea test whilst simultaneously undergoing a sleep study with a Type I sleep monitor (Lab-PSG) and optionally a Type IV sleep monitor.
  Interventions: Device: NightOwl HSAT

INTERVENTIONS:
Device: NightOwl HSAT — Patient wears the NightOwl sensor device

SUMMARY:
Prospective validation study of the NightOwl, a Type IV home sleep apnea test (HSAT), compared to a traditional Type I and a Type IV sleep monitor.

DETAILED DESCRIPTION:
The purpose of this prospective validation study is the evaluation of the accuracy of the NightOwl HSAT to derive parameters relevant for the diagnosis of sleep apnea. The NightOwl HSAT comprises a finger or forehead mounted sensor and an automated analytics software. The sensor measures double-wavelength photo-plethysmography and accelerometry. The analytics software automatically interprets the sensor data and derives a measure of sympathetic activation of the autonomic nervous system, oxygen saturation, instantaneous pulse rate and activity. For each patient in the cohort, the AHI derived by the NightOwl will be compared to that of the Type I sleep monitor (in-lab PSG), which will acquire data simultaneously during the diagnostic night of the patient referred to the sleep lab for a polysomnography. On a randomly selected subset of patients, a Type IV sleep monitor will additionally be applied for comparison of its automated AHI derivation to that of the NightOwl.

ELIGIBILITY:
Inclusion Criteria:

* Indication for a sleep study

Exclusion Criteria:

* Mentally disabled people
* Known allergy to Plexiglas (PMMA) or other acrylates

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 450 (Estimated)
Dates: Start 2017-06-29 (Actual); Primary Completion 2019-09-15 (Estimated); Study Completion 2019-12-15 (Estimated)

PRIMARY OUTCOMES:
Apnea-Hypopnea Index (AHI) | At the time of the diagnostic night
  Comparison of the AHI derived from the NightOwl HSAT to that of the Type I and Type IV sleep monitors

SECONDARY OUTCOMES:
Sleep-wake discrimination | At time of the diagnostic night
  Comparison of the sleep-wake discrimination derived from the NightOwl HSAT to that of the Type I and Type IV sleep monitors

CONTACTS AND LOCATIONS:
Overall Officials: Duarte Mendes de Almeida, Ir., Study Director — Ectosense NV
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Limburg, Belgium

IPD SHARING:
Plan to Share IPD: No